CLINICAL TRIAL: NCT05286125
Title: Erector Spinae Plane Block Versus Oblique Subcostal Transverses Abdominis Plane Block for Controlling Postoperative Pain After Umbilical Hernia Repair
Brief Title: Erector Spinae Plane Block Versus Oblique Subcostal Transverses Abdominis Plane Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Michael Adel Shaker, lecturer of anaesthesia and intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 8034-7-11-2021
Record Dates: First submitted 2021-12-22; First posted 2022-03-18 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Parapsychology; Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erector spinae plane (ESP) block group ( (E) group) (Active Comparator): Under aseptic conditions, a high frequency linear transducer will be placed on the spinous process at T8 level on the parasagittal plane and then slid 2.5-3 cm laterally to visualize the transverse process and erector spinae muscle.
  Interventions: Procedure: erector spinae plane (ESP) block
- oblique subcostal transverse abdominis plane (TAP) block ( (T) group) ) (Active Comparator): Under aseptic conditions, the probe will be initially placed below the xyphoid process to view the linea alba, then directed obliquely down the costal margin while keeping the rectus abdominis muscle in view. The transverse abdominis muscle come into view below the rectus abdominis muscle. The probe will be advanced further until the semilunaris is viewed.
  Interventions: Procedure: oblique subcostal transverse abdominis plane (TAP) block

INTERVENTIONS:
Procedure: erector spinae plane (ESP) block — Using the in plane technique, the needle will be advanced between the transverse process and erector spinae muscle. The correct location will be confirmed using 1ml of Local Anesthetic (LA) to view hydrodissection(12). 19ml of LA will be injected between the muscle and transverse process.
  Arms: erector spinae plane (ESP) block group ( (E) group)
Procedure: oblique subcostal transverse abdominis plane (TAP) block — An echogenic needle will be inserted in-plane until the needle tip reaches the fascia between the rectus abdominis and the transverse abdominis muscles. Once the needle enters the TAP plane, a dynamic injection can be performed by advancing the needle under ultrasound guidance laterally in the pocket created by the initial injection of 5 - 10 mL of local anesthetic; as the needle is advanced, the remaining local anesthetic will be injected. This allows for a more lateral spread of the local anesthetic
  Arms: oblique subcostal transverse abdominis plane (TAP) block ( (T) group) )

SUMMARY:
Comparing the impact of bilateral erector spinae plane block and transverse abdominis plane block on improving quality of pain management after umbilical hernia repair.

DETAILED DESCRIPTION:
Postoperative pain is an important problem after umbilical hernia repair which has negative effects on patient's hemodynamics and cause delayed ambulation resulting in prolonged duration of hospital stay and poor patient satisfaction.

Multiple analgesic strategies have been proposed including Non steroidal anti-inflammatory drugs (NSAIDs), opioids, epidural analgesia. Each of them has its limitations.

Ultra¬sound guided regional anesthesia techniques for abdominal wall can be effective components of multimodal postoperative analgesia with limited side-effects Erector spinae plane (ESP) block is a promising para-spinal bock that can achieve both visceral and somatic abdominal analgesia if the injection was performed at a lower thoracic level. Transverse abdominis plane (TAP) block which is considered a peripheral nerve block that is aimed at anesthetizing nerves supplying the anterior abdominal wall.

We will compare between erector spinae plane block and transverse abdominis plane block for controlling postoperative pain after umbilical hernia repair.

Patients will be allocated randomly into two equal groups by a computer-generated randomization table Group (E) (n=26): Patients will receive erector spinae plane (ESP) block after completion of surgery.

Group (T) (n= 26): Patients will receive oblique subcostal transverse abdominis plane (TAP) block after completion of surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective umbilical hernia repair.
* Patient acceptance.
* Both sex
* Patient's age 21 - 60 years.
* Patients with American Society of Anesthesiologists (ASA) physical status I, II.
* BMI 25 - 30 kg m-2.

Exclusion Criteria:

* Uncooperative patients and patients with psychological problems.
* Patients with liver or renal impairment.
* Patients with contraindication to regional anesthesia.
* Patients with history of allergy to drug used in the study.
* Patients with chronic pain.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesic requirements | 24 hours postoperative
  measuring the total doses of analgesic required to relieve the pain

SECONDARY OUTCOMES:
Postoperative pain severity using Visual Analogue scale | 24 hours postoperative
  assessing pain severity using Visual Analogue scale (VAS) (0-100mm)
Postoperative pain severity using Verbal Rating Scale | 24 hours postoperative
  assessing pain severity using Verbal Rating Scale (mild, moderate and severe)
Postoperative pain severity using Numeric Rating Scale | 24 hours postoperative
  assessing pain severity using Numeric Rating Scale (NRS) (0-10; 0, no pain; 10, worst pain)
Postoperative heart rate changes | 24 hours postoperative
  monitoring postoperative changes in the heart rate (HR) measured by beat per minute (BPM) and comparing it with the preoperative measures
Postoperative blood pressure changes | 24 hours postoperative
  monitoring postoperative changes in the blood pressure (BP) measured by mm Hg and comparing it with the preoperative measures.
Incidence of postoperative side effects | 24 hours postoperative
  recording any postoperative complications as nausea and vomiting
Duration of postoperative hospital stay | 24 hours postoperative
  measuring the delay in discharging the patients postoperative because of the pain

CONTACTS AND LOCATIONS:
Overall Officials: Michael A shaker, lecturer, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University hospital, Zagazig, Sharqia Province, Egypt